CLINICAL TRIAL: NCT00988624
Title: A Phase 1, Randomized, Open-Label, Single Dose Cross-Over Study In Healthy Volunteers To Estimate The Pharmacokinetics Of Four Modified-Release Formulations Of Dimebon (Latrepirdine)
Brief Title: A Study In Healthy Volunteers To Estimate The Pharmacokinetics Of Four Modified-Release Formulations Of Dimebon (Latrepirdine)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B1451023
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Alzheimer's Disease; Huntington Disease
Keywords: bioavailability pharmacokinetics Alzheimer's Disease Huntington Disease
MeSH Terms: conditions — Alzheimer Disease; Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Period 1 (Experimental)
  Interventions: Drug: Dimebon IR Tablet
- Period 2 (Experimental)
  Interventions: Drug: Dimebon MR1
- Period 3 (Experimental)
  Interventions: Drug: Dimebon MR2
- Period 4 (Experimental)
  Interventions: Drug: Dimebon MR3
- Period 5 (Experimental)
  Interventions: Drug: Dimebon MR4

INTERVENTIONS:
Drug: Dimebon IR Tablet — Pharmacokinetics of a single oral dose of 10 mg dimebon immediate release tablet will be assessed on Day 1 - 3.
  Arms: Period 1
Drug: Dimebon MR1 — Pharmacokinetics of a single oral dose of 10 mg dimebon modified release formulation, MR1, will be assessed on Day 1 - 3.
  Arms: Period 2
Drug: Dimebon MR2 — Pharmacokinetics of a single oral dose of 10 mg dimebon modified release formulation, MR2, will be assessed on Day 1 - 3.
  Arms: Period 3
Drug: Dimebon MR3 — Pharmacokinetics of a single oral dose of 10 mg dimebon modified release formulation, MR3, will be assessed on Day 1 - 3.
  Arms: Period 4
Drug: Dimebon MR4 — Pharmacokinetics of a single oral dose of 10 mg dimebon modified release formulation, MR4, will be assessed on Day 1 - 3.
  Arms: Period 5

SUMMARY:
This study will evaluate four different modified release formulation to estimate the amount of dimebon available to the body relative to the current dimebon formulation that is given three times a day. The results of this study will help inform and guide further formulation development efforts with the ultimate goal of reducing dose frequency to once-a-day or twice-a-day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive.

Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subjects with any history of a previous seizure (including childhood febrile seizures) or convulsion or significant head trauma.
* Subjects with hypersensitivity reactions to dimebon or other antihistamines.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* Smokers who use greater than 5 cigarettes per day.
* Use of proton pump inhibitors, antacids, and H2-blockers are prohibited for the duration of the study.
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of non-hormonal contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
PK endpoints for dimebon and M7 (where appropriate) for each formulation: AUC0-24, AUC0-24(dn), AUCinf (as data permit) AUCinf(dn), AUClast, AUClast(dn), Tlag, Cmax, Tmax, and t1/2 (as data permit). | Day 1-3 of Period 1, 2, 3, 4, or 5

SECONDARY OUTCOMES:
Safety and tolerability for each formulation (AEs, ECG, vital signs, safety labs) | Day 1-3 of Period 1, 2, 3, 4, or 5

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1451023&StudyName=A%20Study%20In%20Healthy%20Volunteers%20To%20Estimate%20The%20Pharmacokinetics%20Of%20Four%20Modified-Release%20Formulations%20Of%20Dimebon%20%28Latrepirdine%29